CLINICAL TRIAL: NCT04119648
Title: A Pilot Study of Collaborative Assessment and Management of Suicidality (CAMS-Jobes, 2006; 2016) With Suicidal Children ("CAMS-4Kids")
Brief Title: A Pilot Study of Collaborative Assessment and Management of Suicidality With Suicidal Children ("CAMS-4Kids")
Acronym: CAMS-4Kids
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study ended due to competing clinical demands.
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: The Catholic University of America (Other)
Responsible Party: Principal Investigator, Jeff Bridge, Director, Center for Suicide Prevention and Research, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00793
Record Dates: First submitted 2019-10-07; First posted 2019-10-08 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Suicidal Ideation; Suicide, Attempted
Keywords: Suicide; Child; CAMS
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted; Suicide

STUDY DESIGN:
Intervention Model Description: This study is an open pilot trial of one treatment without control or comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAMS-4Kids (Experimental): Participants will receive up to 10 sessions of CAMS-4Kids
  Interventions: Behavioral: CAMS-4Kids

INTERVENTIONS:
Behavioral: CAMS-4Kids — The Collaborative Assessment and Management of Suicidality (CAMS-Jobes, 2006; 2016) is an evidence-based, therapeutic framework for addressing suicide risk in the adult population. CAMS-4Kids, the research intervention used in this study, is a 10-session developmentally-sensitive adaptation of CAMS for children ages 5 - 11 years old.

SUMMARY:
The purpose of the study is to assess the feasibility and acceptability of CAMS-4Kids for children with suicidal ideation and/or behavior. During this open pilot trial, we will enhance treatment procedures, refine adherence measures, and develop a treatment manual. Our study sample will include 10 children, ages 5 - 11 years old, seeking outpatient services for suicidal ideation and/or behavior.

DETAILED DESCRIPTION:
The Collaborative Assessment and Management of Suicidality (CAMS-Jobes, 2006; 2016) is an evidence-based, therapeutic framework for addressing suicide risk in the adult population. CAMS-4Kids, the research intervention used in this study, is a 10-session developmentally-sensitive adaptation of CAMS for children ages 5 - 11 years old.

Within the CAMS framework, clinicians treat patient-identified issues that contribute to their suicidal thoughts and/or behavior called "suicidal drivers." A "clinical road map" is provided through the Suicide Status Form (SSF) that guides treatment as an assessment, treatment planning, tracking and clinical outcome tool. Clinicians and children engage in the assessment and treatment planning sections of the SSF - Initial Form at the outset of treatment. A CAMS Stabilization Plan is also collaboratively developed which focuses on reducing access to lethal means, coping strategies, decreasing interpersonal isolation, and ways to address potential barriers to care.

Subsequent CAMS-4Kids sessions include ongoing assessment and treatment plan reviews using the SSF - Interim Sessions Form. The CAMS Stabilization Plan is also reviewed and updated as clinically indicated. Treatment involves clinical interventions most appropriate to treat the patient's "suicidal drivers." Clinical interventions may include coping cards, "Hope Journal," behavioral activation, Virtual Hope Box, increasing social support, guided imagery, DBT relaxation skills, positive self-talk, and other cognitive-behavioral techniques.

The conclusion of CAMS-4Kids occurs after 3 consecutive sessions of effectively managing suicidal ideation and behavior. The SSF Outcome/Dispositional Final Session Form is completed at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* children between the ages of 5 - 11 years old, inclusive, at the time of consent;
* current suicidal ideation and/or behavior;
* resides with primary caregiver who has legal authority to consent to research participation
* client of outpatient Behavioral Health Services
* Outpatient or Mood and Anxiety Program visit scheduled at least 4 weeks from the diagnostic assessment and/or discharge from the Crisis Stabilization Unit.

Exclusion Criteria:

* the inability to understand study procedures (e.g. developmental disabilities, severe cognitive impairments, actively psychotic)
* inability of the child and/or parent to speak or read English
* current participation in weekly therapy sessions with outpatient Behavioral Health Crisis Team

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
CAMS-4Kids Suicide Status Form-4 (SSF-4) | Each session measured from baseline up to 12-week follow-up
  The SSF-4 measures overall suicide risk.
Change from baseline in psychosocial functioning and impairment on the Columbia Impairment Scale (CIS) at treatment completion (up to 12 weeks), 3 months and 6 months. | Baseline, Treatment Completion (up to 12 weeks), 3 month and 6 month follow-up
  The CIS is a valid 13-item child- and parent- report measure of psychosocial impairment with good internal consistency and test-retest reliability. Scores range from 0 (no problem) to 4 (very bad problem), with higher scores indicating worse outcomes.
Change from baseline in suicidal ideation and behavior on the Columbia-Suicide Severity Rating Scale (C-SSRS) at treatment completion (up to 12 weeks) 3 months and 6 months | Baseline, Treatment Completion (up to 12 weeks), 3 month and 6 month follow-up
  The C-SSRS is a validated, semi-structured interview that assesses both suicidal behavior and suicidal ideation (yes/no, frequency), with flexible timepoints and multiple informants depending on administrator purpose and need. Scores range 0 (no ideation) to 5 (ideation with plan and intent), with higher numbers indicating worse outcomes. Suicidal behavior is present or absent, presence of behavior indicates worse outcomes.

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | Up to 12-week follow-up
  The CSQ-8 is an 8 item measure of treatment satisfaction with services with both a parent and child version.
Therapeutic Alliance Scale for Children, Revised (TASC-r) | Up to 12-week follow-up
  The TASC-r is a measure of the working child-therapist working relationship.
Therapeutic Alliance Scale for Caregivers and Parents (TASCP) | Up to 12-week follow-up
  The TASCP is a measure of the working caregiver-therapist working relationship.
CAMS Rating Scale | Each session measured from baseline up to 12-week follow-up
  The CAMS Rating scale measures CAMS treatment fidelity.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Bridge, PhD, Principal Investigator — Abigail Wexner Research Institute at NCH
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jobes, D. A. (2016). Managing suicidal risk: A collaborative approach 2nd Ed. New York: Guilford Press.
- [Background] Anderson, A. R., Keyes, G. M. & Jobes, D. A. (2016). Understanding and treating suicidal risk in young children. Practice Innovations, 1(1), 3-19.
- [Background] Comtois KA, Jobes DA, S O'Connor S, Atkins DC, Janis K, E Chessen C, Landes SJ, Holen A, Yuodelis-Flores C. Collaborative assessment and management of suicidality (CAMS): feasibility trial for next-day appointment services. Depress Anxiety. 2011 Nov;28(11):963-72. doi: 10.1002/da.20895. Epub 2011 Sep 21. PMID 21948348
- [Background] Ellis TE, Green KL, Allen JG, Jobes DA, Nadorff MR. Collaborative assessment and management of suicidality in an inpatient setting: results of a pilot study. Psychotherapy (Chic). 2012 Mar;49(1):72-80. doi: 10.1037/a0026746. PMID 22369081
- [Background] Ellis TE, Rufino KA, Allen JG, Fowler JC, Jobes DA. Impact of a Suicide-Specific Intervention within Inpatient Psychiatric Care: The Collaborative Assessment and Management of Suicidality. Suicide Life Threat Behav. 2015 Oct;45(5):556-566. doi: 10.1111/sltb.12151. Epub 2015 Jan 12. PMID 25581595
- [Background] Ellis TE, Rufino KA, Allen JG. A controlled comparison trial of the Collaborative Assessment and Management of Suicidality (CAMS) in an inpatient setting: Outcomes at discharge and six-month follow-up. Psychiatry Res. 2017 Mar;249:252-260. doi: 10.1016/j.psychres.2017.01.032. Epub 2017 Jan 14. PMID 28126581
- [Background] Jobes DA, Wong SA, Conrad AK, Drozd JF, Neal-Walden T. The collaborative assessment and management of suicidality versus treatment as usual: a retrospective study with suicidal outpatients. Suicide Life Threat Behav. 2005 Oct;35(5):483-97. doi: 10.1521/suli.2005.35.5.483. PMID 16268766
- [Background] Ryberg W, Zahl PH, Diep LM, Landro NI, Fosse R. Managing suicidality within specialized care: A randomized controlled trial. J Affect Disord. 2019 Apr 15;249:112-120. doi: 10.1016/j.jad.2019.02.022. Epub 2019 Feb 7. PMID 30771641
- [Background] O'Connor, S. S., Brausch, A. M., Anderson, A. R., & Jobes, D. A. (2014). Applying the Collaborative Assessment and Management of Suicidality (CAMS) to suicidal adolescents. International Journal of Behavioral Consultation and Therapy, 9(3), 53-58.